CLINICAL TRIAL: NCT03211715
Title: Validation of Low Anterior Resection Syndrome Score in Korean Version
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Principal Investigator, Hyung Jin Kim, Assistant Professor, Saint Vincent's Hospital, Korea
Other Study IDs: SVHKorea
Record Dates: First submitted 2017-06-20; First posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Neoplasm of Rectum; Surgery--Complications; Surgery
MeSH Terms: conditions — Rectal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — Rectal cancer patients who received sphincter saving surgery will be asked to fill up questionnaire related to bowel dysfunction

SUMMARY:
In contemporary era of rectal cancer treatment, development of surgical technique and tool, adaptation of chemoradiation therapy, as well as multidisciplinary approach have led increased survival as well as rate of sphincter preservation. However, poor anorectal function, such as fecal incontinence and/or urgency, has also been increased. Such anorectal dysfunction is named as low anterior resection syndrome, and its rate has been reported in 40 to 90% in rectal cancer patients who received sphincter preserving surgery. Low anterior resection syndrome is known to debilitate quality of life in survivors of rectal cancer. Previously, several studies attempted to evaluate the low anterior resection syndrome via questionnaires and scoring system. Adapting the low anterior resection syndrome score system created in Denmark, this study investigates the validity of the scoring system in Korean language.

DETAILED DESCRIPTION:
In this study, the low anterior resection syndrome score questionnaire proposed by Therese Juul is translated to Korean language by 3 different professional translators. Patients who received sphincter saving surgery to treat rectal cancer will be asked to fill up the questionnaire. Compiling the results, the quality of life after sphincter preserving surgery will be investigated in the association with the low anterior resection syndrome.

ELIGIBILITY:
Inclusion Criteria:

* age 20-80
* surgery undertook from Jan. 2009 to Dec. 2016
* diagnosed with adenocarcinoma
* curative intent of surgery
* planned surgery
* sphincter saving surgery

Exclusion Criteria:

* patients with stage IV
* emergency surgery
* patients with recurrent disease

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Rectal cancer patients who underwent sphincter preserving surgery from Jan. 2009 to Dec. 2016 will be included.
  Patients who are in use of stoma despite of preserved sphincter, are with recurrent disease, or in systemic metastasis, who underwent emergency surgery will not be included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-07-19 (Estimated); Primary Completion 2018-07-19 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life in association to the severity of bowel dysfunction | 3 months follow-up, 6 months follow-up, 1 year follow-up, 2 year follow-up, 3 year follow-up, 4 year follow-up, 5 year follow-up, beyond 5 year follow-up
  The change in the quality of life will be evaluated based on the questionnaire in regard to bowel dysfunction

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juul T, Ahlberg M, Biondo S, Espin E, Jimenez LM, Matzel KE, Palmer GJ, Sauermann A, Trenti L, Zhang W, Laurberg S, Christensen P. Low anterior resection syndrome and quality of life: an international multicenter study. Dis Colon Rectum. 2014 May;57(5):585-91. doi: 10.1097/DCR.0000000000000116. PMID 24819098